CLINICAL TRIAL: NCT01928251
Title: Promoting Smoking Cessation in the Community Via Quit to Win Contest 2013: A Prospective Study and a Randomized Controlled Trial
Brief Title: Promoting Smoking Cessation in the Community Via Quit to Win Contest 2013
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. LI William Ho Cheung, Assistant professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QTW2013
Record Dates: First submitted 2013-05-30; First posted 2013-08-23 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Informed early monetary incentive (Experimental): Incentives of abstinence will be given to those who self-report abstinence for the past 7 days at 3-month follow-up and pass the 3-month biochemical validation (Exhaled carbon monoxide level < 4 ppm, saliva cotinine level < 10 ng/ml) (Group A-Q). Participants will be informed about the incentives through telephone follow-up at 1 week and 1 month. Those who have not quitted at 3 months (Group A-N) or those self-reported quitters who refuse to participate in biochemical validation will be informed again that they will be given the same incentive if they have quitted at 6 months and the quitting is validated.
  Interventions: Behavioral: Informed early monetary incentive
- Uninformed early monetary incentive (Experimental): Incentives of abstinence will be given to those who self-report abstinence for the past 7 days and pass the 3-month biochemical validation (Group B-Q), but they will not be informed about the incentive at the 1-week and 1-month follow-up. Those who have not quitted at 3 months (Group B-N) or those self-reported quitters who refuse to participate in the biochemical validation will be informed that they will be given the same incentive if they have quitted at 6 months and the quitting is validated.
  Interventions: Behavioral: Uninformed early monetary incentive
- Uninformed late monetary incentive (No Intervention): Incentives for the self-reported and biochemically-validated abstinence at 6-month follow-up will be given after the 6-month biomedical validation. They would not be informed about the incentive at the 1-week, 1-month and 3-month follow-up. Group C also has two subgroups, those who have quitted at 3 months (Group C-Q) and those who have not (Group C-N).

INTERVENTIONS:
Behavioral: Informed early monetary incentive — Participants will be informed at 1 week after the baseline recruitment about the monetary incentive of quitting.
  Apart from the different arrangement of monetary incentives for the three RCT arms, all participants of the Quit to Win Contest will receive self-help materials on smoking cessation, including a COSH-developed self-help smoking cessation booklet, a health education card, and the quitline (i.e. 1833183). The theory-based health education card (pocket size), which guided by the HAPA, will be developed and distributed to the participants as a reminder and a 'homework assignment' to be completed at home, for the purpose of enhancing their intention and practice of the suggested behaviour (quitting smoking).
  Arms: Informed early monetary incentive
Behavioral: Uninformed early monetary incentive — Participants will be informed at 3 months after the baseline recruitment about the monetary incentive of quitting.
  Apart from the different arrangement of monetary incentives for the three RCT arms, all participants of the Quit to Win Contest will receive self-help materials on smoking cessation, including a COSH-developed self-help smoking cessation booklet, a health education card, and the quitline (i.e. 1833183). The theory-based health education card (pocket size), which guided by the HAPA, will be developed and distributed to the participants as a reminder and a 'homework assignment' to be completed at home, for the purpose of enhancing their intention and practice of the suggested behaviour (quitting smoking).
  Arms: Uninformed early monetary incentive

SUMMARY:
According to the Census & Statistics Department (2011), there are still 659,300 daily smokers (11.1%) in Hong Kong. Smoking and passive smoking kill over 7,000 people per year. Smoking is addictive, and it is difficult for some motivated smokers to quit without assistance. On the other hand, many smokers may not be ready to quit or want to quit on their own, so it is difficult to reach them.

Quit and Win programme is an opportunity to reach and encourage a large group of smokers to make quit attempt. Quit and Win Contest assumes that smokers can develop a higher motivation to quit and gain a wider social support in quitting. According to Cahill and Petera (2011), smokers can develop a high motivation to quit and gain a wider social support through participating in the Quit and Win Contest.

The Hong Kong Council on Smoking and Health (COSH) organized three "Quit to Win Contests" and recruited over 3000 smokers from 2009-2012. These events enhanced the motivation and confidence to quit smoking. Lucky draw was also conducted to attract smokers to quit smoking and winners were validated by biochemical tests.

Community-Based Participatory Research (CBPR) is an partnership approach that can enlighten and utilize the network within communities as community partners can obtain ample manpower and social resources. To effectively raise the awareness of the contest and recruit as many participants as we can from the community, working with NGOs in the 18 Hong Kong districts with a CBPR model may be one effective way of program implementation.

Thus, we proposed to (1) test the effectiveness of combining competition and short-term monetary incentives to motivate smokers who participate in the Quit to Win Contest 2013 to quit smoking; (2) use a Community-Based Participatory Research (CBPR) model to build capacity and to engage community partners in taking on this important public health issue for sustainability in the community; and (3) conduct the process evaluation to assess the effectiveness of the recruitment activity and how it is linked with the overall program outcomes.

Hypothesis:

To examine the effectiveness of the interventions, three arms are (i) Group A: Informed early monetary incentive, which participants will be notified of the incentive through telephone follow-up at 1-week and 1-month follow-ups; (ii) Group B: Uninformed early monetary incentive, which participants will not be informed about the incentive until 3-month telephone follow-up; (iii) Group C (control group): Uninformed late monetary incentive, which participants will not be informed about the incentive throughout 1-week, 1-month and 3-month follow-ups.

The primary outcomes are the self-reported 7-day point prevalence (pp) quit rate at 3 months of group A compared to group B and group C. The secondary outcomes include (i) self-reported 7-day point prevalence (pp) quit rate at 6 months, (ii) biochemical validated quit rates, (iii) rate of smoking reduction by at least half of baseline amount, (iv) number of quit attempts at 3 and 6 months among the three groups and (v) the above cessation outcomes of all subjects, including or not including in the RCT.

DETAILED DESCRIPTION:
According to the report of Census & Statistics Department (Census & Statistics Department (Hong Kong SAR government), 2011), there are still 659,300 daily smokers (11.1%) in Hong Kong. Smoking and passive smoking kills over 7,000 people per year (Lam, Ho, Hedley, Mak, & Peto, 2001). Smoking also led to an annual medical cost, long-term care and productivity loss of US$688 million in 1998 (McGhee et al., 2006), which was equivalent to 0.6% of GDP in the region (Census & Statistics Department (Hong Kong SAR government), 2001). Smoking is addictive, and it is difficult for some motivated smokers to quit without assistance. On the other hand, many smokers may not be ready to quit or want to quit on their own, so it is difficult to reach them.

The Quit and Win programme provides an opportunity to reach and encourage a large group of smokers to make quit attempt, in order to increase the number of quitters. This Quit and Win model assumes that smokers can develop a higher motivation to quit and gain a wider social support in quitting thru participating in this kind of contests (Cahill & Petera, 2011). Such quitting contests or incentive programs appeared to reach a large number of smokers, and demonstrated a significantly higher quit rate for the quit and win group than for the control group (Cahill & Rafael, 2008). Cognitive theory suggested that immediate incentive exerts more influence than delayed reward for implementing more patient preferences (Berns, Laibson, & Loewenstein, 2007). Some critics echoed this by considering to reward the participants who were abstinent or achieved other cessation outcomes in the early stage of the quitting process, instead of a later cessation outcome (Aveyard & Bauld, 2011). Among the three overseas studies attempted to combine short-term monetary reward and competition as the incentive for abstinence (Glasgow, Hollis, Ary, & Boles, 1993; Hennrikus, Jeffery, Lando, & Murray, 2002; Koffman, Lee, Hopp, & Emont, 1998), Koffman's study in the workplace supported that participants with short-term incentives had a higher quit rate at 6 months than others without the incentives.

In 2009, we conducted a 3-armed randomized controlled trial to compare the effectiveness of two additional interventions of a 3-minute brief telephone advice and 8 mobile phone messages to the usual care of smoking cessation self-help material in the Quit to Win Contest 2009 (Chan, 2011). More than one thousand participants were successfully recruited in a period of one and half months, with an overall self-reported quit rate of 21.6% among the contestants. However, the additional brief telephone advice or the SMS messages did not show a higher quit rate than control group. In 2010, we conducted another RCT on the Quit to Win Contest 2010 to compare the effectiveness of an on-site face-to-face brief smoking cessation advice versus self-help materials (control) on quit rate and changes in smoking behaviors. Once again, we recruited over one thousand participants during a period of 2.5 months. A higher quit rate was observed in the intervention group (18.4%), in which participants received an on-site brief counselling, than the control group (13.8%) at 6-month follow-up, although it was marginally statistically insignificant (p = 0.08) (Wong & Chan, 2012). In 2012, the RCT in the Quit to Win Contest tested the effectiveness of the on-site counselling with telephone boosters and health education card theoretically based on the Health Action Process Approach for the intervention group (Schwarzer, 2008). HAPA suggests that one's intention of behaviour change can be fostered by knowing that the new behaviour has positive outcomes as opposed to the negative outcomes that accompany the current behaviour; and planning (action planning and coping planning) serves as an operative mediator between intentions and behaviour. In addition, another SMS intervention group received 16 SMS about cessation advice and motivation within one month. The quit rates for these two intervention groups were 9.4% and 11.5%, respectively, but they did not differ from the control group significantly (9.7%).

The three Quit to Win Contests in Hong Kong recruited over 3,000 smokers from the community who otherwise might not even think about quitting smoking. On the other hand, the engagement in the competition boosted up the confidence and motivation to quit among smokers who joined the Quit to Win contest, but additional counselling and short messaging services did not increase the quit rate. All the three contests conducted a lucky draw to select a few prize winners whose abstinence was validated by biochemical tests. In accordance with the research direction suggested by the above foreign studies, the forthcoming RCT on Quit to Win Contest will explore the effectiveness of short-term monetary incentives combined with the prizes of the lucky draws.

Community-Based Participatory Research (CBPR) is a partnership approach in a scientific research that involves the collaboration among community partners and academic researchers throughout the research process (Israel, Schulz, & Parker, 1998). It has been found effective in enhancing community input, building community capacity, and addressing barriers to health in study participants who have historically been underrepresented in research (Andrews, Newman, Heath, Williams, & Tingen, 2012; Horowitz, Robinson, & Seifer, 2009). Community partners have the capability of mobilizing local social resources and manpower, and utilizing their network within the community, which are beneficial to a scientific research involving population-based interventions. To effectively raise the awareness of the contest and recruit as many participants as we can from the community, working with NGOs in the 18 Hong Kong districts with a CBPR model may be one effective way of program implementation.

The challenge of applying the CBPR model in the smoking cessation program is to equip the staff from NGOs and HKU about the related skills and knowledge, and maintain the quality of research process and intervention. Process evaluation is a systematic procedure during the delivery of public health interventions in order to understand how well the program does and to link the progress to outcomes (Centers for Disease Control and Prevention, 2008). In addition to the training programme and briefing session to be provided to the participating NGOs, monitoring and documentation are needed throughout the recruitment and research process so that the quality and integrity of the effort by the involved NGOs can be evaluated.

To conclude, we proposed to (1) test the effectiveness of combining competition and short-term monetary incentives to motivate smokers who participate in the Quit to Win Contest 2013 to quit smoking; (2) use a Community-Based Participatory Research (CBPR) model to build capacity and to engage community partners in taking on this important public health issue for sustainability in the community; and (3) conduct the process evaluation to assess the effectiveness of the recruitment activity and how it is linked with the overall program outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged 18 or above
* Smoke at least 1 cigarette per day in the past 3 months
* Able to communicate in Cantonese
* Exhaled carbon monoxide (CO) 4 ppm or above, assessed by a validated CO smokerlyzer

Exclusion Criteria:

* Smokers who have difficulties (either physical or cognitive condition) to communicate
* Currently following other smoking cessation programs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1143 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Self-reported quit rate | 3 months after recruitment
  Self-reported 7-day point prevalence quit rate after 3 months

SECONDARY OUTCOMES:
Biochemically validated and self-reported smoking habit at 3 and 6 months | 3 and 6 months after recruitment
  (i) self-reported 7-day point prevalence (pp) quit rate at 6 months, (ii) biochemical validated quit rates, (iii) rate of smoking reduction by at least half of baseline amount, (iv) number of quit attempts at 3 and 6 months among the three groups and (v) the above cessation outcomes of all subjects, including or not including in the RCT.

CONTACTS AND LOCATIONS:
Overall Officials: William Li, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong SAR, China